CLINICAL TRIAL: NCT02166619
Title: Transcranial Direct Current Stimulation in Rehabilitation of Chronic Stroke Patients: Multicenter Clinical Trial
Brief Title: tDCS in Poststroke on Upper Limb Rehabilitation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Kátia Monte-Silva, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChronicStroke_tDCS_rehab
Record Dates: First submitted 2014-06-14; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-05

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; Electric stimulation therapy; Neuroplasticity
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tDCS + physical therapy (Experimental): Firstly, patients will undergo electrophysiological evaluation: motor evoked potential, motor threshold and silent period in both hemispheres. After those procedures, bihemispheric tDCS will be applied with duration of 20 minutes, intensity of 2 mA where anodal electrode will be on the affected hemisphere and the cathodal electrode, on the non-affected hemisphere. After tDCS, patients will be submitted to 40 minutes of physical therapy protocol. Experimental sessions will be repeated five times per week to complete 10 sessions.
  Interventions: Device: tDCS + physical therapy
- Sham tDCS + physical therapy (Sham Comparator): Firstly, patients will undergo electrophysiological evaluation: motor evoked potential, motor threshold and silent period in both hemispheres. After those procedures, bihemispheric sham tDCS will be applied. Anodal electrode will be on the affected hemisphere and the cathodal electrode, on the non-affected hemisphere. Sham tDCS will be performed by ramping current flow for the first 10 seconds of stimulation, but switching the stimulator off after 30 seconds. After bihemispheric sham tDCS, patients will be submitted to 40 minutes of physical therapy protocol. Experimental sessions will be repeated five times per week to complete 10 sessions.
  Interventions: Device: tDCS + physical therapy

INTERVENTIONS:
Device: tDCS + physical therapy — Bihemispheric tDCS involves application of very low-amplitude direct currents (2 mA or less) via surface scalp electrodes. It produces a sub-sensory level of electrical stimulation wich remains imperceptible by most people during application. In a small percentage of patients, it may cause minimal discomfort with a mild tingling sensation, which usually disappears after a few seconds. Depending on the polarity, tDCS can increase or decrease corticomotor excitability. Anodal tDCS is able to facilitate neurons depolarization - increasing cortical excitability - while, on the other hand, cathodal tDCS hyperpolarizes the resting membrane potential, reducing the neuronal firing and the cortical excitability.
  Other: Physical Therapy
  Other Names: non invasive brain stimulation, neuroConn (Germany)

SUMMARY:
In this study, the investigators wondered whether bihemispheric transcranial direct current stimulation (tDCS) would be capable to potentialize the effects of physical therapy on upper limb rehabilitation of chronic stroke patients. Moreover, the study aims to investigate the pattern of physiological variables involved in the recovery of these patients. For this purpose, patients included will be submitted to 10 sessions with active or sham bihemispheric tDCS associated with intensive and individual physical therapy session.

DETAILED DESCRIPTION:
Patients will undergo behavioral and electrophysiological evaluation before, immediately after, 30 and 90 days after 10 sessions (follow ups). They will be submitted to the following evaluations: (i) Fugl-Meyer Scale; (ii) Jebsen-Taylor hand functional test; (iii) Box-Block test; (iv) Motor Activity Log - 30; (v) Geriatric Depression Scale - 15; (vi) Beck Depression Inventory; (vii) Stroke Impact Scale; (viii) Hand Grip Strength and (iv) Modified Ashworth Scale. In addition, one question of motivation will be answered by patients in different stages of the treatment: (i) motivation regarding their own life at the beginning and ending of the treatment; (ii) daily motivation at the beginning of each session; (iii) motivation of the last week at the fifth and tenth sessions; (iv) motivation regarding their own life at 30 and 90 days after the ending of the treatment. A visual scale will be used to assess patient's motivation through five potential answers: "very little", "little", "more or less", "very much" and "extremely".

Electrophysiological measures will be performed before and after each session and in follow ups.

Evaluation of brain activity will be performed using single-pulse transcranial magnetic stimulation (TMS-p) only in Recife Centre. Magnetic stimulation (Neurosoft, Russia) will be applied through a figure-8 coil to determine motor cortex representation of first dorsal interosseus muscle (hotspot) and performed the following electrophysiological measures, in both cerebral hemispheres, to assess cortical activity: (i) Motor Evoked Potential (MEP); (ii) Active motor threshold (AMT) and (iii) Silent period (PS).

Evaluation of brain activity will be performed using single-pulse transcranial magnetic stimulation (TMS-p) only in Recife Centre. Magnetic stimulation (Neurosoft, Russia) will be applied through a figure-8 coil kept at a 45 degree angle relative to the sagittal line and pointed to the anterior region of the skull. Firstly, patients will be instructed to sit in a chair and to search a comfortable position. TMS-p will be applied in both motor cortex, healthy and injured, to determine the cortical representation of first dorsal interosseus muscle. The hotspot will be considered the most excitable area, with more intense motor evoked potential (MEP), measured by electromyography.

The following electrophysiological measures will be performed in both cerebral hemispheres to assess cortical activity:

(i) Motor Evoked Potential (MEP) : the intensity of magnetic stimulator is adjusted to produce an average MEP of 1.0 mV. TMS-p will be applied in the area of cortical representation of the first dorsal interosseous and mean responses to stimuli should reach 0.8 mV to 1.2 mV.

(ii) Active motor threshold (AMT) : will be request to the patient to perform contraction of the first interosseous muscle and then, will be given ten pulses by TMS-p to determinate active motor threshold. Motor threshold corresponds to the lowest intensity of TMS-p to produce a MEP of 50 μV in 50% of the pulses applied to the hotspot.

(iii) Silent period (PS) : is the interval of time that usually is observed absence of electromyographic activity. Occurs immediately after the registration of MEP during voluntary contraction of the target muscle (PEMvc - motor evoked potentials recorded during voluntary contraction). Higher the intensity of the magnetic stimulation, longer the duration of PS.

During tDCS application, patients will be seated in a comfortable chair with head and arms rests. Current will be applied by a DC stimulator (NeuroConn, Germany) using a pair of saline-soaked sponge electrodes (surface 24 cm²).

Bihemispheric tDCS will be applied to primary motor cortex (M1) in left and right hemispheres. These points correspond to C3 and C4 according to International 10-20 EEG system. Anode will be placed to M1 in affected hemisphere, while the cathode is positioned to M1 over the unaffected hemisphere. Parameters of current intensity and duration (dose) used were previously established in poststroke patients: 2 mA stimulation intensity for 20 minutes with current ramping up and down of 10 seconds each.

Sham tDCS has been used in several studies to evaluate the effect of active tDCS. In placebo stimulation, intensity and electrode's positions are the same as in the active group, however, current duration is only 30 seconds, with current ramping up and down of 10 seconds each. Moreover, the electrostimulation device is automatically turned off without patient's perception. Thus, patients experience early sensations (mild to moderate tingling) in stimulation site without inducing effect. Moreover, after each tDCS session, patients will answer adverse effects questionnaire.

After apply tDCS, 40 minutes of individual and intensive physical therapy session will be performed. Goals of the physical therapy protocol were discussed based in neuroplasticity principles by a group of experienced physiotherapists. Physical therapy activities will be focused on rehabilitation of upper limb and will cover the following purposes: flexibility, transfer and posture, coordination, balance and sensorial stimulation. Depending on patient's ability, a program of activities for each purpose will be adapted by a trained physical therapist.

The study will be conducted simultaneously in three research centers in Brazil: Applied Neuroscience Laboratory (LANA), Universidade Federal de Pernambuco (UFPE), Pernambuco, Brazil; D'Or Institute for Research and Education (ID'Or), Botafogo, Rio de Janeiro, Brazil and at the University Center Augusto Mota (UNISUAM), Bonsucesso Unit, Rio de Janeiro, Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Primary or recurrent, ischemic or hemorrhagic stroke, confirmed by computed tomography or magnetic resonance imaging
* Chronic Stroke (> 12 months)
* Sensorimotor sequelae in an upper limb due to stroke
* Score ≥ 18 at Folstein Mini Mental State Examination
* Score ≥ 4 at Ashworth Scale
* Minimal active wrist movement (flexion and extension)
* At least one pinch movement

Exclusion Criteria:

* Prior neurological diseases
* Multiple brain lesions
* Metal implant in the skull and face
* Pacemaker
* History of seizures
* Epilepsy
* Pregnancy
* Hemodynamic instability
* Performing physical therapy elsewhere during the period of intervention
* Score > 59 at the Fugl-Meyer Assessment of Motor Recovery after Stroke
* Traumatic or orthopedic lesion limiting the range of motion of upper limb

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer assessment of paretic upper limb motor function | baseline, after sessions, 30 and 90 days
  Fugl-Meyer assessment is used to measure motor control recovery. It is a 226-point scoring system that includes the following sessions: range of motion, pain, sensation, motor function of upper and lower limbs, balance and coordination/velocity. We will apply only two sessions: upper limb motor function and coordination/velocity. These sessions totalize 66 points.The instrument provides a reliable and valid measure of specific motor function that is also sensitive to change.

SECONDARY OUTCOMES:
Change from Motor Activity Log-30 | baseline, after sessions, 30 and 90 days
  MAL is a scripted, structured interview to measure real-world upper extremity function. It was developed to measure the effects of therapy on the most impaired arm following stroke. Consists of 30 activities of daily living such as using a towel, brushing teeth and picking up a glass. For a specified time period post-stroke, patients are asked about the extent of activity performance and how well it was performed by the most impaired arm. Response scale ranges from 0 (never used) to 5 (same as pre-stroke). Scores average for activity frequency comprises the Amount of use scale (AOU); the mean of scores for how well the activity was performed comprises Quality of movement (QOM). Ideally, ratings are obtained from patient and as well as the caregiver.

OTHER OUTCOMES:
Change from Jebsen-Taylor Hand Function Test | baseline, after sessions, 30 and 90 days
  Jebsen-Taylor Hand Function Test was designed to provide short, objective test of hand functions commonly used in daily living activities. Targeted patient population included adults with neurological and musculoskeletal conditions involving hand disabilities, although there may be other patient populations with other hand dysfunction which may be appropriate. The test was developed to be used by health professionals working in restoration of hand function. It consists of seven items that includes a range of fine motor, weighted and unweighted hand function activities.

CONTACTS AND LOCATIONS:
Overall Officials: Kátia Monte-Silva, PhD, Study Director — Applied Neuroscience Laboratory, Universidade Federal de Pernambuco
Locations (3):
- Brazil (3):
  - Applied Neuroscience Laboratory, Universidade Federal de Pernambuco, Recife, Pernambuco
  - D'Or Institute for Research and Education (ID'Or), Rio de Janeiro, Rio de Janeiro
  - University Center Augusto Mota (UNISUAM), Rio de Janeiro, Rio de Janeiro

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411